CLINICAL TRIAL: NCT00312234
Title: Feasibility and Impact of Qigong as Compared to Aerobic Exercise in the Treatment of Childhood Chronic Musculoskeletal Pain: A Pilot Randomized Controlled Trial.
Brief Title: Qigong vs. Aerobic Exercise in the Treatment of Childhood Chronic Musculoskeletal Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Brian Feldman, Division Head, Rheumatology, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000007434
Record Dates: First submitted 2006-04-05; First posted 2006-04-07 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Muscular Disease; Fibromyalgia
Keywords: Muscular Disease; Fibromyalgia; Exercise Therapy; Qigong; Aerobic Exercise; pediatrics
MeSH Terms: conditions — Muscular Diseases; Fibromyalgia | interventions — Exercise

INTERVENTIONS:
Behavioral: Aerobic exercise
Behavioral: Qigong exercise

SUMMARY:
This study is comparing two different exercise programs, Qi Gong (gentle stretching, and breathing) with an aerobics program (boxing and dancing) to see if children with chronic pain or fibromyalgia are able to take part in the program. We would also like to know if it is easy to take part in an exercise program.

We hypothesize that children with chronic musculoskeletal pain and FM, who engage in Qigong fitness training, will be more compliant, and have an equivalent or possibly superior improvement on measures of motor function (peak power, endurance, and metabolic efficiency) compared to children given an aerobic fitness exercise program.

DETAILED DESCRIPTION:
Background: Childhood fibromyalgia (FM) and chronic musculoskeletal pain are common and sometimes devastating pediatric disorders resulting in widespread pain, fatigue, tenderness and significant disability. Exercises, including vigorous aerobics, and complementary and alternative health strategies - like Qigong - have shown to be safe and effective in the treatment of adult FM and chronic pain. Qigong may be more tolerable than more vigorous exercise. No data is available for this treatment in children.

Research Question: To test the feasibility of studying Qigong exercise versus aerobic fitness exercise to reduce symptoms and disability in children with FM or chronic pain.

Methods: Randomized single-blind pilot study of 30 childhood FM/chronic pain patients allocated to either 12 weeks of supervised Qigong therapy or 12 weeks of supervised graded aerobic exercise training (cardio-karate).

Expected Results: Physical exercise training - whether Qigong or aerobic exercise - represents a potentially feasible, safe and effective alternative therapy and may increase the ability for these children to resume their normal activities of daily life. Exercise training may therefore emerge as a pivotal mode of therapy for all children with FM/chronic pain. Results from our study will allow us to plan a definitive study.

Specific Objectives: 1. To study the feasibility of enrolling, randomizing and studying participants with FM/chronic pain using validated measures of symptoms, physical and psychosocial function, quality of life and exercise testing. 2. Acquire pilot data that will allow for the estimation of an effect size for the comparison of 2 forms of exercise - standard aerobic fitness exercise, and a specially designed Qigong program. This effect size estimate will be used in designing a subsequent definitive randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-18 years
* Diagnosis of childhood fibromyalgia or chronic musculoskeletal pain (ACR criteria)

Exclusion Criteria:

* Co-morbidity with cardiac, pulmonary or metabolic disease.
* Children who engage in more than 3 hours of structured extracurricular physical activity programs weekly, unless a physiotherapy pool program with emphasis on joint range of motion and stretching.
* Children who are unable to cooperate with testing procedures.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30
Dates: Start 2005-08; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Accrual rates
Compliance with therapy
Acceptability of exercise program
Degree of conditioning of subjects at baseline
Proportion of completed exercise tests and questionnaires
Dropout rates
Estimates of the effect sizes for exercise tests and questionnaire data

CONTACTS AND LOCATIONS:
Overall Officials: Brian Feldman, MSc MD FRCPC, Principal Investigator — The Hospital for Sick Children
Locations (2):
- Canada (2):
  - Bloorview MacMillan Children's Centre, Toronto, Ontario
  - Hospital for Sick Children, Toronto, Ontario

REFERENCES:
- [Derived] Stephens S, Feldman BM, Bradley N, Schneiderman J, Wright V, Singh-Grewal D, Lefebvre A, Benseler SM, Cameron B, Laxer R, O'Brien C, Schneider R, Silverman E, Spiegel L, Stinson J, Tyrrell PN, Whitney K, Tse SM. Feasibility and effectiveness of an aerobic exercise program in children with fibromyalgia: results of a randomized controlled pilot trial. Arthritis Rheum. 2008 Oct 15;59(10):1399-406. doi: 10.1002/art.24115. PMID 18821656